CLINICAL TRIAL: NCT01852981
Title: Evaluation Study of Interventions for Physical Activity Promotion in Primary Health Care/Health Family Strategy in Brazil.
Brief Title: Evaluation Study of Interventions for Physical Activity Promotion in Primary Health Care in Brazil.
Acronym: PACTIVEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Alex Antonio Florindo, Ph.D., University of Sao Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2009/14119-4; NCT01330836 (obsolete NCT alias)
Record Dates: First submitted 2010-10-19; First posted 2013-05-14 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: Physical Activity
Keywords: Physical activity promotion; Intervention; Public Health
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Lifestyle counseling (Experimental): Physical activity promotion using methods based on health education.
  Interventions: Behavioral: Lifestyle counseling
- Supervised exercise (Experimental): Supervised sessions of aerobic, strength, and stretching exercises, drawn up in accordance to the American College of Sports Medicine recommendations.
  Interventions: Behavioral: Supervised exercise
- Control (No Intervention): Control group.

INTERVENTIONS:
Behavioral: Lifestyle counseling — Strategies consisted of group discussion, some physical activities, phone support, and printed materials. The content and strategies were elaborated by a team formed by a doctor, nutritionists, a psychologist, and physical education professionals and the main aim was to promote the engagement in physical activity, working not only on behavioral change but also on the environment attributes available for physical activity practice. The main strategy was the group discussion, which sessions lasted 120 minutes each and its frequency changed as follow: in the first month they were weekly; in the second occurred twice per month; and in the third month onwards sessions were monthly. All sessions occurred in the Primary Health Unit or inside a community association building.
  Arms: Lifestyle counseling
Behavioral: Supervised exercise — Supervised exercise program in groups. Individuals in this program participated in three weekly structured and supervised sessions of aerobic, strength, and stretching exercises, drawn up in accordance to the American College of Sports Medicine recommendations. Load, intensity, and exercise adjustments were made during the program. All sessions lasted 60 minutes each and occurred in a gymnasium nearby the Primary Health Unit.
  Arms: Supervised exercise

SUMMARY:
To verify changes in physical activity levels, metabolic markers, and physical fitness as results of two physical activity interventions within the Brazilian public health system (primary health care).

DETAILED DESCRIPTION:
The effects of two strategies - lifestyle counseling focused on physical activity, and supervised exercise - adapted to the Brazilian primary health care system and resources will be compared between them and with a control group. Subjects are healthy, physically inactive adults from a low socioeconomic area of Sao Paulo city. Evaluations will be done at the study baseline, 6 months, 12 months, and 18 months (6 months follow-up) after the beginning. The primary outcome is leisure-time physical activity.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or more;
* To be registered in the Brazilian public health system.

Exclusion Criteria:

* Practice of leisure-time physical activity in the previous month;
* Practice of transport-related physical activity (walking or cycling) for at least 150 minutes in the previous week;
* Diagnostic of type II diabetes or severe arterial hypertension;
* Use of beta-blockers for treating hypertension or cardiovascular disease;
* Health problem or disease that would make the individual incapable of leaving home and making the journey to practice physical activity;
* Diseases such as cancer, cirrhosis, chronic kidney disease, chronic obstructive pulmonary disease osteoporosis and severe depression at advanced stages;
* Cognitive problem or disease that would not allow the individual from answering the questionnaire alone;
* Being morbidly obese, with a body mass index (BMI) ≥40 kg/m2;
* To have plans to move house over the two-year subsequent period;
* Being pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2011-02; Primary Completion 2012-02 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline leisure-time physical activity at 12 months | 12 months
Change from baseline leisure-time physical activity at 18 months | 18 months

SECONDARY OUTCOMES:
Change from baseline leisure-time physical activity at 6 months | 6 months
Change from baseline transport-related physical activity at 12 months | 12 months
Change from baseline transport-related physical activity at 6 months | 6 months
Change from baseline transport-related physical activity at 18 months | 18 months
Change from baseline quality of life at 12 months | 12 months
Change from baseline quality of life at 18 months | 18 months
Change from baseline physical fitness at 12 months | 12 months
Change from baseline physical fitness at 18 months | 18 months
Change from baseline body composition at 12 months | 12 months
Change from baseline body composition at 18 months | 18 months
Change from baseline blood pressure at 12 months | 12 months
Change from baseline blood pressure at 18 months | 18 months
Change from baseline blood glucose at 12 months | 12 months
Change from baseline blood glucose at 18 months | 18 months
Change from baseline blood lipids at 12 months | 12 months
Change from baseline blood lipids at 18 months | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Alex A Florindo, Ph.D., Principal Investigator — University of Sao Paulo
Locations (2):
- Brazil (2):
  - University of Sao Paulo, São Paulo, São Paulo
  - School of Arts, Sciences and Humanities, University of Sao Paulo, São Paulo, São Paulo

REFERENCES:
- [Derived] Salvador EP, Ribeiro EH, Garcia LM, Andrade DR, Guimaraes VM, Aoki MS, Florindo AA. Interventions for physical activity promotion applied to the primary healthcare settings for people living in regions of low socioeconomic level: study protocol for a non-randomized controlled trial. Arch Public Health. 2014 Mar 13;72(1):8. doi: 10.1186/2049-3258-72-8. PMID 24624930
- See also: Research group website. — http://www.each.usp.br/gepaf